CLINICAL TRIAL: NCT02537691
Title: A Prospective, Single Arm, Longitudinal Cohort Study To Assess Biomarkers In Real World Patients With Severe Asthma
Brief Title: Longitudinal Cohort Study in Participants With Severe Asthma to Assess Biomarkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MB29599; 2015-000742-35 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Theophylline; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled Corticosteroids (ICS) + Controller Medications (Other): Participants with severe asthma Global Initiative for Asthma (GINA) step 4/5 as indicated by current treatment with daily ICS consisting of >/=500 mcg FP administered by DPI (or equivalent), and at least one of the following controller medications: LABAs, LTRAs, LAMAs, theophylline or oral corticosteroids.
  Interventions: Drug: FP; Drug: LABA; Drug: LTRA; Drug: LAMA; Drug: Theophylline; Drug: Oral Corticosteroids

INTERVENTIONS:
Drug: FP — ICS consisting of FP will be administered by DPI (or equivalent) as per investigator discretion.
Drug: LABA — LABA will be administered as per investigator discretion.
Drug: LTRA — LTRA will be administered as per investigator discretion.
Drug: LAMA — LAMA will be administered as per investigator discretion.
Drug: Theophylline — Theophylline will be administered as per investigator discretion.
Drug: Oral Corticosteroids — Oral corticosteroids will be administered as per investigator discretion.

SUMMARY:
Prospective, single-arm, longitudinal, international, multicenter study in a real-world cohort of adult severe asthma participants being conducted to assess the relationships between asthma biomarkers and asthma-related health-outcomes for a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed by a respiratory physician greater than or equal to (>/=) 12 months prior to study enrolment
* Pre-bronchodilator FEV1 of 30 percent (%) to 85% at baseline/Visit 1
* Documented bronchodilator response defined as >/=12% relative improvement in FEV1 after bronchodilator administration or a positive methacholine bronchial challenge test with provocative concentration causing a 20% fall in FEV1 (PC20) less than (<) 8 milligrams (mg) at study baseline/Visit 1 or within 24 months prior to baseline
* Current treatment with a total daily dose of >/= 500 micrograms (mcg) of fluticasone propionate (FP) dry powder inhaler (DPI) (or equivalent ) and at least one of the following controller medications: long-acting Beta-agonist (LABA), leukotriene receptor antagonist (LTRA), long-acting muscarinic antagonists (LAMAs), theophylline or oral corticosteroids, with a continued duration of three months prior to baseline/Visit 1

Exclusion Criteria:

* Acute or chronic parasitic, bacterial, fungal or viral infections that required, or currently require, hospitalization or antimicrobial treatment during the last four weeks prior to participant eligibility
* Acute asthma exacerbation or any other medical event treated with increased doses of oral, or any dose of intramuscular (IM) or intravenous (IV) corticosteroids within six weeks prior to study
* Other relevant pulmonary diseases (e.g. chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis) requiring treatment within 12 months prior to baseline/Visit 1
* Ex-smokers with >/=10 pack-year smoking history
* Prior treatment with bronchial thermoplasty
* Participation in any clinical trial of an investigational agent or procedure within six months prior to baseline/Visit 1 or during the study
* Pregnancy prior to participation or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Mean Number of Asthma Exacerbations in Participants With High Baseline Periostin Compared to participants With Low Baseline Periostin | Baseline up to Week 52

SECONDARY OUTCOMES:
Percentage of Participants With Asthma Exacerbations | Baseline up to Week 52
Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Specified Time Points | Baseline, Weeks 26, 52
Time Taken for the Occurrence of First Asthma Exacerbation | Baseline up to Week 52
Time to Treatment Failure | Baseline up to Week 52
Change From Baseline in Mini Standardized Asthma Quality of Life Questionnaire (MiniAQLQ) at Specified Time Points | Baseline, Weeks 13, 26, 39, 52
Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) at Specified Time Points | Baseline, Weeks 13, 26, 39, 52 or within 12 weeks of last visit for early termination (up to Week 52)
Change From Baseline in Asthma Control Test (ACT) at Specified Time Points | Baseline, Weeks 13, 26, 39, 52 or within 12 weeks of last visit for early termination (up to Week 52)
Percentage of Participants With Changes to Standard of Care (SoC) Asthma Treatment as Reported by the Investigator and Confirmed by Study Steering Committee | Baseline up to Week 52
Serum Periostin Levels During the Study | Baseline, Weeks 26, 52
Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) Levels | Baseline, Weeks 26, 52
Blood Eosinophil Levels During the Study | Baseline, Weeks 26, 52
Serum Immunoglobulin E (IgE) Levels During the Study | Baseline, Weeks 26, 52
Number of Urgent Asthma-Related Health Care Utilization: Hospitalizations | Weeks 13, 26, 39, 52
Number of Urgent Asthma-Related Health Care Utilization: Emergency Department Visits | Weeks 13, 26, 39, 52
Number of Urgent Asthma-Related Health Care Utilization: Acute Care Visits | Weeks 13, 26, 39, 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (100):
- United States (29):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Southern California Research Center, Mission Viejo, California
  - Capital Allergy Resp Dis Ctr, Sacramento, California
  - Allergy Assoc Medical Group, San Diego, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - AAADRS; Clinical Research Center, Coral Gables, Florida
  - Volunteer Medical Research, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Albany, Georgia
  - Asthma & Allergy Center, P.C., Papillion, Nebraska
  - Allergy & Asthma Research of Nj, Inc, Mount Laurel, New Jersey
  - Island Medical Research Pc, Commack, New York
  - Winthrop University Hospital, Mineola, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Vital Prospects Clin Res Pc, Tulsa, Oklahoma
  - Allergy-Asthma Specialists PC, Blue Bell, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allergy & Clinical Immun Assoc, Pittsburgh, Pennsylvania
  - Berks-Schuylkill Respiratory Specialists, Ltd, Wyomissing, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Allergy & Asthma Res Ctr PA, San Antonio, Texas
  - Allergy Associates of Utah, Murray, Utah
  - Bridgerland Clinical Research, North Logan, Utah
  - Northridge Internal Medicine, Charlottesville, Virginia
  - O & O Alpan, LLC, Fairfax, Virginia
  - ASTHMA, Inc, Seattle, Washington
  - Pulmonary & Sleep Research, Spokane, Washington
- Belgium (5):
  - Hospital Erasme; Neurologie, Brussels
  - Private Practice, Jambes
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - CHU UCL Mont-Godinne, Mont-godinne
- Bulgaria (2):
  - Mhat - Pleven; Clinic of Pulmonology, Pleven
  - Specialized Hospital for Active Treatment for pneumo-phtysiatric diseases, Rousse
- Canada (8):
  - Vancouver General Hosp; The Lung Centre, Vancouver, British Columbia
  - St. Paul's Hospital University of British Colambia Division of Hematology, Vancouver, British Columbia
  - Burlington Lung Clinic, Burlington, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital; Endoscopy Department, Montreal, Quebec
  - Hopital Laval; Centre de Pneumologie, Québec
- Denmark (2):
  - Hvidovre Hospital, Lungemedicinsk Afdeling, Hvidovre
  - Lungemedicinsk afd. L, Bispebjerg Hospital, København NV
- Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris, France
- Germany (9):
  - Institut für Allergie- und Asthmaforschung Berlin, IAAB, Berlin
  - Berufsgenossenschaftliches Uni-Klinikum Bergmannsheil GmbH, Bochum
  - Lungenzentrum Darmstadt, Darmstadt
  - Ruhrlandklinik Lungenzentrum der UNI Essen Abt.Pneumologie-Allergologie, Essen
  - Universitätsklinikum Freiburg, Abteilung Pneumologie, Freiburg im Breisgau
  - Pneumologicum, Hanover
  - KPPK Studienzentrum GmbH; Dr. med. A. Kroker, Dr. med. O. Schmidt, Koblenz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Medizinische Klinik, Pneumologie, Mainz
  - Klinikum der Universität München; Campus Großhadern; Med. Klinik und Poliklinik V, München
- Hungary (5):
  - Dr. Kenessey Albert Korhaz Es Rendelointezet; Tudoosztaly (Pulmonolgy Dept ), Balassagyarmat
  - Synexus Magyarorszag Kft, Budapest
  - Szent János Kórház; Tüdőgondozó Intézet és Szűrőállomás, Budapest
  - Debrecen Uni Medical School; Dept of Pulmonary Medicine, Debrecen
  - Matrai Állami Gyógyintézet ; Bronchológia, Mátraháza
- Italy (7):
  - Presidio Ospedaliero SS. Annunziata di Chieti ; Dip. Medico-UOSD Allergologia, Chieti, Abruzzo
  - Policlinico di Modena; Oncologia, Ematologia e Patologie dell'apparato Respiratorio, Modena, Emilia-Romagna
  - IRCCS AOU SAN MARTINO - IST;UO ALLERGOLOGIA-IMMUNOPATOLOGIA RESPIRATORIA e TERAPIE BIOTECNOLOGICHE, Genoa, Liguria
  - AOU Città della Salute e della Scienza di Torino - Ospedale Le Molinette; SC Pneumologia, Turin, Piedmont
  - Azienda Policlinico Vittorio Emanuele; Pneumologia Riabilitativa E Allergologia, Catania, Sicily
  - A.O. Ospedali Riuniti; Villa Sofia-Cervello di Palermo; U. O. Pneumologia 2 - Padiglione B, Palermo, Sicily
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
- Latvia (3):
  - Clinical Hospital Gailezers; Dept of Pulmonology, Riga
  - Riga 1st hospital, outpatient clinic Bruninieks, Riga
  - Latvian University postgraduate institute, Riga
- Netherlands (3):
  - Spaarne Ziekenhuis Hoofddorp; Long Geneeskunde, Hoofddorp
  - Medisch Centrum Leeuwarden; Longziekten, Leeuwarden
  - St. Antonius; R&D Long, Nieuwegein
- CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia, Portugal
- Russia (9):
  - Research Institute of Complex Cardiovascular Pathology, Kemerovo
  - SBIH "Clinical dermatovenerologic dispensary " of Ministry of Health of the Krasnodar region, Krasnodar
  - FSBI "National Research Center - Institute of Immunology" of FMBA of Russia, Moscow
  - SBEI APE Russian Medical Academy of Post-graduate Education; Department of Clinical Allergology, Moscow
  - SBHI of NN region "RCH of NN n.a. N.A.Semashko", Nizhny Novgorod
  - City Hospital #40 of Resort Administrative District, Saint Petersburg
  - City Out-patient Clinic #106, Saint Petersburg
  - Saratov State Medical University; Chair Of Clinical Allergology, Saratov
  - SBEI HPE "North Ossetian State Medical Academy" of Ministry of Health of Russia, Vladikavkaz
- Spain (7):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, LA Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda; Servicio de Neumología, Majadahonda, Madrid
  - Hospital de Galdakano; Servicio de Neumologia, Galdakano, Vizcaya
  - Fundacio Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I provincial; Servicio de Neumologia, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Neumología, Córdoba
  - Hospital Universitario 12 de Octubre; Servicio de Neumologia, Madrid
- United Kingdom (9):
  - Queen Elizabeth Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Gloucestershire Royal Hospital, Gloucester
  - William Harvey Research Institute, London
  - St George's Hospital, London
  - North Manchester Hospital; Respiratory Department, Manchester
  - Freeman Hospital; Respiratory Department; Sir William Leach Lung Research Centre, Newcastle upon Tyne
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Royal Shrewsbury Hospital, Shrewsbury